CLINICAL TRIAL: NCT02298465
Title: Randomized Controlled Study on Extracorporeal Shockwave Lithotripsy for Distal Ureteric Stone: Transgluteal Versus Traditional Prone Approach
Brief Title: ESWL for Distal Ureteric Stone: Supine Versus Prone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Ho, Resident Specialist (Urology), Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QueenMaryH
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Urinary Tract Stones; Urinary Stones; Urinary Calculi
Keywords: ESWL; distal ureteric stone; transgluteal; supine ESWL
MeSH Terms: conditions — Urinary Calculi | interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prone ESWL (Active Comparator): ESWL for distal ureteric stone is performed in the traditional prone position
  Interventions: Procedure: Prone ESWL; Device: Extracorporeal Shockwave Lithotripsy (ESWL)
- Supine ESWL (Experimental): ESWL for distal ureteric stone is performed in the supine position, with the shockwave generator head placed at a 30 degree angle to the vertical at the patient's gluteal muscles. Thus, the shockwaves will travel via the greater and lesser sciatic foramina to reach the stone
  Interventions: Procedure: Supine ESWL; Device: Extracorporeal Shockwave Lithotripsy (ESWL)

INTERVENTIONS:
Procedure: Supine ESWL — ESWL to distal ureteric stone is performed in the supine position with the shockwave generator placed in the patient's buttock area. The aim is to direct the shockwaves through the greater and lesser sciatic foramina to reach the distal ureter.
  Arms: Supine ESWL
Procedure: Prone ESWL — ESWL to the distal ureteric stone is performed in the traditional prone position. The shockwave generator is placed on the patient's abdomen
  Other Names: Transgluteal
  Arms: Prone ESWL
Device: Extracorporeal Shockwave Lithotripsy (ESWL) — The ESWL machine we use is the Dornier S2 lithotriptor. ESWL is performed without any sedation or anesthesia under fluoroscopy. Painkillers are given upon request.

SUMMARY:
Extracorporeal shockwave lithotripsy (ESWL) for urinary stone is common and widespread nowadays. Approximately 80% of urinary stones are treated by ESWL. Traditionally distal ureteric stones are treated with ESWL in the prone position. However, as some patients cannot tolerate lying in the prone due to medical illness such as chronic obstructive pulmonary disease (COPD), some authors have reported using the supine approach of ESWL for treatment of distal ureter stones. No serious complications had developed in the patients who underwent supine approach. Only minor complications such as self-limiting blood in the urine, painful passage of urine, or local pain that had responded to oral painkillers. There were no serious complications encountered in children as well. In the most recent retrospective review by Tolley et al, they had revealed that patients who had underwent supine ESWL for distal ureteric stones had an improved stone-free rate compared with the traditional prone approach.

Patient with radio-opaque distal ureteric stones (stones below the sacroiliac joint) on KUB X-ray, who have opted for ESWL treatment, are randomized into two groups: one undergoing ESWL in the supine position and the other undergoing ESWL in the prone position. Patients will be observed for two hours after ESWL before being discharged. Oral painkillers as necessary will be provided to the patient. The patients will have a KUB Xray at 2 weeks post-ESWL, and then monthly afterwards if required. If there are residual stones at the 2-week follow-up, the patient will be offered ESWL again. Patients are free to withdraw from the study at any time and will continue to be managed as per usual.

The investigators aim to have 130 patients, with 65 patients in each group with an interim analyses to be performed when 66 patients have been recruited (33 patients in each group).

DETAILED DESCRIPTION:
Previous authors have reported using the greater and lesser sciatic foramina as a pathway for the shockwaves to reach the distal ureter. No serious complications had developed in the patients who underwent transgluteal approach. Only minor complications such as self-limiting hematuria, dysuria, or pain that had responded to oral analgesics. There were no serious complications encountered in children as well. In the most recent retrospective review by Tolley et al, they had revealed that patients who had underwent transgluteal ESWL for distal ureteric stones had an improved stone-free rate of 78% in the transgluteal group versus 40% in the prone group after one session of shockwave lithotripsy and a stone-free rate of 92% versus 63% respectively after two sessions of shockwave lithotripsy. This has been speculated to be due to the presence of bowel gas attenuating the shockwaves as well as a long skin-to-stone distance in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* All patients, over 18 years of age, with distal ureteric stones with stone size of ≥3mm on kidney-ureter-bladder (KUB) X-ray who opted for ESWL treatment

Exclusion Criteria:

* Patients who are unable to provide consent
* radiolucent stones
* active urinary tract infections
* pregnancy
* uncontrolled hypertension
* uncontrolled bleeding tendencies
* severe skeletal malformations
* arterial aneurysms within the vicinity of the stone (such as iliac artery aneurysms)
* unable to assume the appropriate position (prone or supine) for ESWL
* solitary kidneys
* transplanted kidneys
* presence of ureteric stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | 2 weeks. If stone still present, then 6 weeks and 10 weeks.
  To review KUB to determine if distal ureteric stone have been passed

SECONDARY OUTCOMES:
Complications rates concerning the two approaches of ESWL | 2 weeks. If stone still present, then 6 weeks and 10 weeks.
  To see if any complications arise from the procedures
Pain associated with the procedure for the two approaches of ESWL | 2 weeks. If stone still present, then 6 weeks and 10 weeks.
  * Using visual analogue scale to determine the pain scores of each intervention on the day of intervention
  * Number of tablets of analgesics used in-between follow up

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ho, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins AD, Gillenwater JY. Extracorporeal shock wave lithotripsy in the prone position: treatment of stones in the distal ureter or anomalous kidney. J Urol. 1988 May;139(5):911-5. doi: 10.1016/s0022-5347(17)42713-3. PMID 3361661
- [Background] Zehntner CH, Marth D, Zingg EJ. ESWL treatment with ventral shock-wave application: therapy of iliac and distal ureteral calculi. Urology. 1991 Jul;38(1):51-3. doi: 10.1016/0090-4295(91)80013-w. PMID 1866859
- [Background] Lu J, Sun X, He L. Sciaticum majus foramen and sciaticum minus foramen as the path of SWL in the supine position to treat distal ureteral stone. Urol Res. 2010 Dec;38(6):417-20. doi: 10.1007/s00240-010-0285-2. Epub 2010 Jul 13. PMID 20625895
- [Background] Sun X, He L, Lu J, Cong X, Shen L, Wang Y, Zhu H. Greater and lesser ischiadic foramina as path of shock wave lithotripsy for distal ureteral stone in children. J Urol. 2010 Aug;184(2):665-8. doi: 10.1016/j.juro.2010.03.060. Epub 2010 Jun 19. PMID 20639031
- [Background] Phipps S, Stephenson C, Tolley D. Extracorporeal shockwave lithotripsy to distal ureteric stones: the transgluteal approach significantly increases stone-free rates. BJU Int. 2013 Jul;112(2):E129-33. doi: 10.1111/j.1464-410X.2012.11738.x. Epub 2013 Jan 29. PMID 23360696